CLINICAL TRIAL: NCT06033599
Title: Motivational Interviewing (MI) and Mindfulness-Oriented Recovery Enhancement (MORE) for Tobacco Dependence and Other Drug Use in Methadone Treatment
Brief Title: Motivational Interviewing and Mindfulness-Oriented Recovery Enhancement
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University of Utah (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nina A. Cooperman, Psy. D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2022001551; R01DA057631 (NIH)
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Polysubstance Abuse; Opioid Use; Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — Nicotine Replacement Therapy; Self-Help Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- MORE and MI (Experimental)
  Interventions: Other: MORE and MI and NRT
- MORE and No MI (Experimental)
  Interventions: Other: MORE and No MI and NRT
- Support Group and MI (Active Comparator)
  Interventions: Other: Support Group and MI and NRT
- Support Group and No MI (Active Comparator)
  Interventions: Other: Support Group and No MI and NRT

INTERVENTIONS:
Other: MORE and MI and NRT — Eight group Mindfulness Oriented Recovery Enhancement sessions and one motivational interviewing session and nicotine replacement therapy.
  Arms: MORE and MI
Other: MORE and No MI and NRT — Eight group Mindfulness Oriented Recovery Enhancement sessions and nicotine replacement therapy.
  Arms: MORE and No MI
Other: Support Group and MI and NRT — Eight group support group sessions and one motivational interviewing session and nicotine replacement therapy.
  Arms: Support Group and MI
Other: Support Group and No MI and NRT — Eight group support group sessions and and nicotine replacement therapy.
  Arms: Support Group and No MI

SUMMARY:
The purpose of this study is to 1) examine barriers and facilitators to implementation of MI and MORE for polysubstance use and evaluate strategies for optimizing training, fidelity, and clinic uptake, and 2) evaluate patient outcomes related to the effectiveness of MORE decreasing opioid, tobacco, and other drug use.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age ≥18
* Currently on methadone; and 4) currently smoke cigarettes.

Exclusion Criteria:

* Severe cognitive impairment (score >23 on Mini Mental Status Exam) or psychosis (positive SCID Psychotic Screen)
* Suicidal risk (score ≥7 on Suicidal Behaviors Questionnaire)
* Inability to attend or fully participate in intervention sessions or assessments
* Previous formal mindfulness training (e.g., MBSR, MBRP) or MORE (from the R21 or R33
* Currently taking smoking cessation pharmacotherapy or participating in smoking cessation counseling
* Any contraindications for NRT
* Currently or soon planning to be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Days of Drug Use | Baseline through 52 weeks.
  Number of days of drug use as measured by self-reported days of use and biochemically verified use via drug screen.
Days of Tobacco Use | Baseline through 52 weeks.
  Number of days of tobacco use as measured by self-reported days of use and biochemically verified use via expired carbon monoxide.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Cooperman, PsyD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (2):
- United States (2):
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
All participant individual data will be available after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available three months through five years after study publication
Access Criteria: Researchers who provide a methodologically sound proposal.